CLINICAL TRIAL: NCT04036383
Title: Effects of Different Type Exercise Trainings on Functionality in Older Fallers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayşe Abit Kocaman (Other)
Responsible Party: Sponsor-Investigator, Ayşe Abit Kocaman, Research Assistant, Kırıkkale University
Organization: Kırıkkale University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FALL AND SQUARE STEP EXERCİSE
Record Dates: First submitted 2019-07-12; First posted 2019-07-29 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Fall Patients

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- vestibüler (Active Comparator): vestibular exercise training
  Interventions: Other: vestibular exercise training; Other: Balance training with computerized balance system; Other: square step exercises
- balance training (Experimental): vestibular exercise training+ balance training with computerized balance system
  Interventions: Other: vestibular exercise training; Other: Balance training with computerized balance system; Other: square step exercises
- square-step (Experimental): vestibular exercise training+ square step exercise
  Interventions: Other: vestibular exercise training; Other: Balance training with computerized balance system; Other: square step exercises

INTERVENTIONS:
Other: vestibular exercise training — The home exercise program consists of vestibulookular reflex stimulating exercises, lower extremity somatosensory system training, static and dynamic balance exercises
Other: Balance training with computerized balance system — Thanks to the receivers under the Neurocom balance master platform, the data of the center of gravity is transferred to the system and visual feedback is provided. Qualitative information reflects progression during static and dynamic postural exercises of the patient. To correct the load distribution, it is necessary to move the cursor to the specified targets in the exercises. The degree of difficulty of training can be increased by increasing the distance between the targets, reducing the time required to reach the targets, changing foot positions or adding upper extremity activity.
Other: square step exercises — Elderly individuals in the square step exercise group will perform step exercises on 2.5x1.0 m thin cushions divided into 40 equal parts. Square step exercises include exercises that include anterior, posterior, lateral and diagonal directions of increasing difficulty. The order of the training program is at four different levels and is organized according to small, basic, regular and advanced levels.

SUMMARY:
The aim of this study to examine the effectiveness of different types of exercise trainings on functionality in older faller

DETAILED DESCRIPTION:
Individuals participating in the study will be blinded and 30 elderly individuals will be included. Sociodemographic information of individuals, Mini Mental State Test, Fall Efficacy Scale, Dynamic Gait Index, Montreal Cognitive Assessment Scale, Daily Life Activities Scale for Vestibular Disorders, World Health Organization Quality of Life Scale-Elderly Module test results will be recorded. Hip flexors and abductors, m.quadriceps femoris and m.tibialis anterior muscle strength will be measured by manual muscle dynamometer. In balance assessments; sensory organization test and adaptation test of computerized dynamic posturography will be recorded. Individuals will be divided into 3 groups by blocking and stratification randomization method. All individuals in the group will perform vestibular exercise training twice a day for 8 weeks as a home exercise program. In the first group, vestibular exercise training will be used as a home program, in the second group, individual rehabilitation program will be applied to the computerized balance system and in the third group, square step exercises will be applied. Exercise training will be held 3 times a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older individuals,
* Mini Mental State Examination Test score above 24,
* At least two falls in the last year
* Independent individuals in mobilization without walking aid

Exclusion Criteria:

* Cardiac diseases
* Pulmonary embolism and deep vein thrombosis in the last three months,
* A history of cerebral aneurysm or intracranial hemorrhage,
* Acute retinal hemorrhage or previous ophthalmic surgery,
* Active infection,
* Multiple organ failure,
* Terminal disease status,
* A history of fractures in the lower and upper extremities within the last three months,
* Severe hearing and vision loss,
* Patients with Alzheimer's disease, Parkinson's disease, dementia
* Patients diagnosed with Benign Paroxysmal Positional Vertigo,
* Those who have received exercise training in the last 6 months,

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Balance Function Assessment-Sensory Organization Test | 5 minutes
  Sensory Organization Test (SOT): This is a six-part test that objectively identifies abnormalities in somatosensory, visual, and vestibular systems that provide postural control.
  The result is a ratio between 0-100 and 100 means perfect stability.
Cognitive Function assessment | 10 minutes
  Cognitive function will be assessed with "Montreal Cognitive Assessment Scale(MoCA)"The MoCA is a screening instrument that evaluates cognitive domains on a single page and scores range from 0 to 30."0" points indicate poor cognitive functions, "30" points indicate good cognitive functions. Increase in scores indicates better cognitive functions.
Gait Function assessment | 15 minutes
  Dynamic Gait Index will be used to evaluate the adaptations during the patient's gait. It evaluates activities such as slow walking, fast walking, walking with head movements, turning, stepping up, jumping obstacles, 0 points are weak and 3 points are successful. Low scores from the scale are indicative of disorders that may cause falls.A total of 8 parameters are evaluated over 24 points.
Balance Function Assessment- Adaptation Test | 5 minutes
  Adaptation Test (ADT):This test evaluates the patient's response to sudden changes and irregularities in the ground and the ability to reduce oscillations. The oscillation energy score is obtained by measuring the force applied to the force platform for recovery. Scores between 0 and 200.Since the maximum score given by the device is 200, the score of that test is considered as 200 in case of a fall. The oscillation energy score is close to 0, indicating better postural adaptation.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe ABİT KOCAMAN, Principal Investigator — Kırıkkale University
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)

REFERENCES:
- [Background] Duque G, Boersma D, Loza-Diaz G, Hassan S, Suarez H, Geisinger D, Suriyaarachchi P, Sharma A, Demontiero O. Effects of balance training using a virtual-reality system in older fallers. Clin Interv Aging. 2013;8:257-63. doi: 10.2147/CIA.S41453. Epub 2013 Feb 28. PMID 23467506
- [Background] Shigematsu R, Okura T, Nakagaichi M, Tanaka K, Sakai T, Kitazumi S, Rantanen T. Square-stepping exercise and fall risk factors in older adults: a single-blind, randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2008 Jan;63(1):76-82. doi: 10.1093/gerona/63.1.76. PMID 18245764
- [Background] Shigematsu R, Okura T, Sakai T, Rantanen T. Square-stepping exercise versus strength and balance training for fall risk factors. Aging Clin Exp Res. 2008 Feb;20(1):19-24. doi: 10.1007/BF03324743. PMID 18283224
- [Background] Fisseha B, Janakiraman B, Yitayeh A, Ravichandran H. Effect of square stepping exercise for older adults to prevent fall and injury related to fall: systematic review and meta-analysis of current evidences. J Exerc Rehabil. 2017 Feb 28;13(1):23-29. doi: 10.12965/jer.1734924.462. eCollection 2017 Feb. PMID 28349029
- [Background] Moreira Bittar RS, Simoceli L, Bovino Pedalini ME, Bottino MA. The treatment of diseases related to balance disorders in the elderly and the effectiveness of vestibular rehabilitation. Braz J Otorhinolaryngol. 2007 May-Jun;73(3):295-8. doi: 10.1016/s1808-8694(15)30071-9. PMID 17684648